CLINICAL TRIAL: NCT01008605
Title: Representative Users Study Of Operating Characteristics Of The Caverject Delivery System.
Brief Title: Caverject User Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A6711035
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2012-03-28 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caverject Impulse (Experimental): representative users
  Interventions: Other: delivery system

INTERVENTIONS:
Other: delivery system — syringe

SUMMARY:
The purpose of this study is to demonstrate the usability of the system.

DETAILED DESCRIPTION:
demonstrate usability

ELIGIBILITY:
Inclusion Criteria:

Age 40 to 70

Exclusion Criteria:

Prior syringe skills

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6711035&StudyName=Caverject%20user%20study

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants who delivered a predefined dose and volume of Alprostadil (prostaglandin E1 [PGE1], Caverject) into a receptacle, using the assigned Caverject Impulse delivery system. Participants did not receive study medication and were monitored during the handling of the Caverject Impulse delivery system.
Period: Overall Study
Arm/Group | All Participants
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 51.6 (8.5)
Age, Customized [Number; unit: participants]
  Between 18 and 44 years | 11
  Between 45 and 64 years | 31
  >= 65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Successfully Operated the Caverject Impulse Delivery System
Description: Percentage of participants who were able to successfully expel the selected dose from the Caverject Impulse Delivery System when relying on the modified Instructions for Use. The process was considered successful if the lower bound of the 95% confidence interval (CI) was more than (>) 80% overall.
Time Frame: Day 1
Population: Full Analysis Set (FAS): All eligible participants who read the instructions and attempted to deliver Alprostadil using the Caverject Impulse Delivery System. Each participant tested one device/dose combination.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
percentage of participants | 95.83
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; Lower limit, 95% one-sided CI = 95.83, 95% CI 1-sided [lower limit 87.46]

2. Secondary Outcome: Number of Participants With Categorical Responses to the Participant Assessment Tool: Question 1
Description: Participant Assessment Tool, Question 1: Instructions provided were useful? Participant responses were reported as follows: Very Useful, Somewhat Useful, Not Very Useful, Not Useful At All.
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
participants
  Very useful | 44
  Somewhat useful | 4
  Not very useful | 0
  Not useful at all | 0

3. Secondary Outcome: Number of Participants With Categorical Responses to the Participant Assessment Tool: Question 2
Description: Participant Assessment Tool, Question 2: Instructions provided were clear? Participant responses were reported as follows: Very Clear, Somewhat Clear, Not Very Clear, Not Clear At All.
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
participants
  Very clear | 43
  Somewhat clear | 4
  Not very clear | 1
  Not clear at all | 0

4. Secondary Outcome: Number of Participants With Categorical Responses to the Participant Assessment Tool: Question 3
Description: Participant Assessment Tool, Question 3: Most difficult step? Participant responses were reported as follows: No Steps Particularly Difficult, Attaching Needle, Mixing Solution, Getting The Air Out Of Syringe, Dialing Dose, Pushing Plunger, Other.
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
participants
  No steps particularly difficult | 38
  Attaching needle | 2
  Mixing solution | 1
  Getting the air out of syringe | 0
  Dialing dose | 2
  Pushing plunger | 4
  Other | 1

5. Secondary Outcome: Number of Participants With Categorical Responses to the Participant Assessment Tool: Question 4
Description: Participant Assessment Tool, Question 4: Syringe easy to use? Participant responses were reported as follows: Very Easy, Somewhat Easy, Somewhat Difficult, Very Difficult
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 48
participants
  Very easy | 43
  Somewhat easy | 4
  Somewhat difficult | 1
  Very difficult | 0

6. Secondary Outcome: Time Required to Perform Each Step While Using the Caverject Impulse Delivery System
Description: Steps involved while using the Caverject Impulse Delivery System included assembly, mixing the dose, de-aeration, setting the dose, and injecting the dose.
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination. n = number of participants with available data.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Caverject 10 Mcg Device, 2.5 Mcg Dose Setting: Participants used the 10 microgram (mcg) Caverject Impulse Delivery System to expel Alprostadil 2.5 mcg in a receptacle. Participants did not receive study medication.
- Caverject 10 Mcg Device, 5.0 Mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Delivery System to expel Alprostadil 5.0 mcg in a receptacle. Participants did not receive study medication.
- Caverject 10 Mcg Device, 7.5 Mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Delivery System to expel Alprostadil 7.5 mcg in a receptacle. Participants did not receive study medication.
- Caverject 10 Mcg Device, 10 Mcg Dose Setting: Participants used the 10 mcg Caverject Impulse Delivery System to expel Alprostadil 10.0 mcg in a receptacle. Participants did not receive study medication.
- Caverject 20 Mcg Device, 5.0 Mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Delivery System to expel Alprostadil 5.0 mcg in a receptacle. Participants did not receive study medication.
- Caverject 20 Mcg Device, 10.0 Mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Delivery System to expel Alprostadil 10.0 mcg in a receptacle. Participants did not receive study medication.
- Caverject 20 Mcg Device, 15.0 Mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Delivery System to expel Alprostadil 15.0 mcg in a receptacle. Participants did not receive study medication.
- Caverject 20 Mcg Device, 20.0 Mcg Dose Setting: Participants used the 20 mcg Caverject Impulse Delivery System to expel Alprostadil 20.0 mcg in a receptacle. Participants did not receive study medication.
Arm/Group | Caverject 10 Mcg Device, 2.5 Mcg Dose Setting | Caverject 10 Mcg Device, 5.0 Mcg Dose Setting | Caverject 10 Mcg Device, 7.5 Mcg Dose Setting | Caverject 10 Mcg Device, 10 Mcg Dose Setting | Caverject 20 Mcg Device, 5.0 Mcg Dose Setting | Caverject 20 Mcg Device, 10.0 Mcg Dose Setting | Caverject 20 Mcg Device, 15.0 Mcg Dose Setting | Caverject 20 Mcg Device, 20.0 Mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 6
seconds
  Step 1: Assembly (n=6, 6, 6, 7, 6, 5, 6, 6) | 103.2 (16.98) | 141.7 (26.17) | 119.2 (58.60) | 115.4 (33.53) | 127.5 (54.57) | 110.2 (31.40) | 109.7 (28.77) | 107.2 (52.70)
  Step 2: Mixing solution (n=6, 5, 6, 7, 5, 5, 6, 6) | 55.5 (28.28) | 57.4 (30.94) | 61.0 (38.78) | 58.0 (37.1) | 50.2 (22.97) | 43.8 (38.21) | 61.2 (16.44) | 51.8 (35.31)
  Step 3: De-aerating (n=6, 5, 6, 7, 5, 5, 6, 6) | 55.8 (18.27) | 50.8 (18.2) | 62.3 (41.55) | 52.7 (26.02) | 48.8 (43.00) | 44.0 (18.12) | 48.2 (18.18) | 57.2 (20.18)
  Step 4: Setting the dose (n=6, 4, 6, 7, 5, 5, 6, 6 | 21.0 (9.65) | 24.8 (7.09) | 70.3 (106.57) | 47.3 (37.80) | 43.2 (41.76) | 26.2 (14.60) | 23.8 (11.37) | 37.3 (22.34)
  Step 5: Injecting dose (n=6, 5, 6, 7, 5, 5, 6, 6) | 98.7 (85.41) | 39.2 (21.21) | 62.8 (68.99) | 80.0 (85.65) | 42.0 (28.55) | 51.6 (42.69) | 31.0 (14.34) | 41.5 (18.22)

7. Secondary Outcome: Number of Participants Providing Comments to Any Question on the Participant Assessment Tool
Description: Number of participants providing comments on questions in the Participant Assessment Tool. Questions were as follows: were instructions clear, were instructions useful, which was the most difficult step, and was the syringe easy to use.
Time Frame: Day 1
Population: FAS. Each participant tested one device/dose combination.
Measure: Number; unit: participants
Arm/Group | Caverject 10 Mcg Device, 2.5 Mcg Dose Setting | Caverject 10 Mcg Device, 5.0 Mcg Dose Setting | Caverject 10 Mcg Device, 7.5 Mcg Dose Setting | Caverject 10 Mcg Device, 10 Mcg Dose Setting | Caverject 20 Mcg Device, 5.0 Mcg Dose Setting | Caverject 20 Mcg Device, 10.0 Mcg Dose Setting | Caverject 20 Mcg Device, 15.0 Mcg Dose Setting | Caverject 20 Mcg Device, 20.0 Mcg Dose Setting
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 6 | 5 | 6 | 6
participants
  Instructions provided were useful? | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
  Instructions provided were clear? | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Most difficult step? | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 2
  Syringe easy to use? | 1 | 2 | 2 | 1 | 2 | 0 | 0 | 2

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.